CLINICAL TRIAL: NCT04613726
Title: Intravenous Granisetron Provides Less Ephedrine Requirement Than Ondansetron in Patients Undergoing Cesarean Section With Spinal Anesthesia: A Randomised Placebo-controlled Trial
Brief Title: The Effect of Intravenous Granisetron and Ondansetron in Patients Undergoing Cesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet AKSOY, Assoc. Prof. Dr. Mehmet AKSOY, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B.30.2.ATA.0.01.00/166
Record Dates: First submitted 2020-10-23; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Vomiting, Postoperative; Postoperative Complications; Hypotension
Keywords: cesarean section; granisetron; ondansetron; spinal anesthesia; blood pressure; pre-treatment
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Postoperative Complications; Hypotension | interventions — Ondansetron; Granisetron; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Comparator / control treatment Control group consisted of patients receiving IV 10 ml normal saline. A comparator group consisted of receiving IV 8 mg ondansetron diluted in 10 ml of normal saline, Another comparator group consisted of receivingIV 3 mg granisetron diluted in 10 ml of normal saline.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist in charge, and the patient and investigators were blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IV 10 ml normal saline (Placebo Comparator): Control group consisted of patients receiving IV 10 ml normal saline.
  Interventions: Drug: Saline
- IV 8 mg ondansetron in 10 ml of normal saline (Active Comparator): This group consisted of receiving IV 8 mg ondansetron diluted in 10 ml of normal saline,
  Interventions: Drug: ondansetron
- IV 3 mg granisetron in 10 ml of normal saline (Active Comparator): This group consisted of receiving IV 3 mg granisetron diluted in 10 ml of normal saline.
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: ondansetron — group consisted of receiving IV 8 mg ondansetron diluted in 10 ml of normal saline
  Arms: IV 8 mg ondansetron in 10 ml of normal saline
Drug: Granisetron — Another comparator group consisted of receivingIV 3 mg granisetron diluted in 10 ml of normal saline
  Arms: IV 3 mg granisetron in 10 ml of normal saline
Drug: Saline — Control group consisted of patients receiving IV 10 ml normal saline
  Arms: IV 10 ml normal saline

SUMMARY:
This study compared the effects of prophylactic intravenous (IV) infusion of ondansetron and granisetron before the spinal anesthesia on hemodynamic parameters in patients undergoing elective cesarean section.

DETAILED DESCRIPTION:
A total of 120 parturients who agreed to participate in the study with uncomplicated term pregnancy, aged between 18-45 years, American society of anesthesiologist I or II undergoing elective cesarean section with combined spinal-epidural anesthesia (CSEA) were included. Participants with complicated pregnancy such as diabetes, pregnancy-induced hypertension or chronic hypertension, fetal anomaly, a history of allergy to study drugs, psychiatric diseases, coagulation abnormalities and mul¬tiple pregnancies were excluded from the study. Also, patients receiving selective serotonin reuptake inhibitors were excluded.

A day before surgery, detailed anamnesis was obtained from the patients and a general systemic examination was performed. Also, patients were informed about the study protocol and written informed consent was obtained. The patients were informed that they should be fasting for 8 hours before surgery. On the day of operation, peripheral intravenous (IV) access was provided using a 16-gauge/18-gauge cannula.

After all patients received 500 ml of Ringer Lactate as preload, they were transferred to the operating room. None of the patients received premedication. Before the anesthesia procedure; patients' age, weight, height, ASA physical status, baseline systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) were recorded. The study medications were prepared by an anesthesia resident who was not involved in the study. Three groups (n=40, for each group) were formed by randomization using a computer-generated table of random numbers. The anesthesiologist in charge, and the patient and investigators were blinded to the group allocation.

Five minutes before the CSEA procedure, Group I received IV 8 mg ondansetron diluted in 10 ml of normal saline, Group II received IV 3 mg granisetron diluted in 10 ml of normal saline, and Group III received IV 10 ml normal saline. Subsequently, combined spinal-epidural anesthesia (CSEA) in the sitting position was performed in all patients. Following skin sterilization and local anesthetic infiltration (2% lidocaine), 18 gauge Tuohy needle (Set for CSEA, Braun®, Melsungen, Germany) was advanced through the midline L2-3 or L3-4 intervertebral spaces with loss of resistance technique. A 27-gauge pencil point needle was inserted intrathecally, using the needle-through-needle technique. After free cerebrospinal fluid flow was observed, 1.8 ml 0.5% isobaric bupivacaine (9 mg) and 15 µg fentanyl was administered over 30 seconds. Then, the spinal needle was removed and epidural catheter was advanced 3 to 5 cm into the epidural space. The catheter was secured in place after it was checked with negative pressure. At the end of the anesthesia procedure, patients were placed in the supine position for operation and the operating table was tilted 20° to the left. Sensory block level was evaluated via pinprick test and when the sensory block reached at the upper level of T6 dermatome, surgery was initiated. If sensory block were not observed within the first 20 min following the spinal injection, spinal anesthesia was considered as failed. In this instance, additional 5 ml solution of 2% lidocaine was injected via the epidural catheter until a T6 level of the sensory block was provided and these patients were excluded from the study. Motor block level was evaluated with Modified Bromage scale (scale 0 = The patient is able to move hip, knee, ankle, and toes.; scale 1 = The patient is able to the full flexion of foot and knee, she is unable to hip flexion; scale 2 = The patient is able to the full flexion of foot, she is unable to knee and hip flexion; scale 3 = Total motor block is available). General anaesthesia protocol was planned in case of three unsuccessful attempts to reach to intrathecal space. Oxygen was delivered during surgery. Intravenous ephedrine (6 mg) was planned to treat hypotension (a 30% decrease in systolic blood pressure compared to preoperative values) and intra¬venous atropine (1 mg) was planned in case of bradycardia (the heart rate < 45 beats/minute) during surgery. In case of nausea and vomiting, intravenous metoclopramide (10 mg) was administered. Following drug administration to the intrathecal space, intraoperative hemodynamic changes were recorded every 2 min for 20 min and then every five minutes until the end of the operation by an anesthetist who was blinded to the group allocation. The operation time (the time from the beginning of the surgical incision until the end of surgery), anesthetic complications such as pruritus and nausea-vomiting and the number of patients requiring epidural medication, ephedrine and atropine during surgery were recorded. Neonatal Apgar scores at 1 and 5 min after delivery and umbilical artery blood gas values were recorded.

After operation, patients were evaluated in the recovery room for 120 min. Visual analogue scale (VAS, 0 cm= no pain, 10 cm= worst pain) scores for pain severity, anesthesia-related side effects (e.g., nausea, vomiting and headache), sensory block time (from the spinal injection to the recovery of T10 dermatome), and the time requiring supplemental analgesics was recorded by an independent observer blinded to the group assignment at 30 min and 1st and 2nd hours post-operatively. In the case of VAS > 3 in a patient, 10 ml solution of 0.1% bupivacaine was given via the epidural catheter. Patients were transferred to the ward, following the motor block had regressed to the T10 level.

The primary end point of the study was the ephedrine requirement during surgery. The minimum sample size required for this study was calculated using the Russ Lenth's Power and sample size calculation application. Thirty-five patients in each group were needed to demonstrate a mean difference in the requirement of 10 mg ephedrine among groups with a power of 90% and alpha 5%. However, a sample size was determined as 40 in each group, considering potential dropouts.

Data were expressed as mean values ± standard deviation (SD) or number and percentage values. Comparisons were performed using the ANOVA test. The percentage values were compared using chi-square, P<0.05 was considered significant statistically.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-45 years
* uncomplicated term pregnancy
* ASA (American society of anesthesiologist) I or II
* undergoing elective cesarean section with combined spinal-epidural anesthesia

Exclusion Criteria:

* psychiatric diseases
* preeclampsia
* pregnancy-induced hypertension
* chronic hypertension
* diabetes
* multiple pregnancies
* fetal anomaly
* allergy to study drugs
* receiving selective serotonin reuptake inhibitors

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with uncomplicated term pregnancy
Enrollment: 120 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
ephedrine requirement | Every two minutes during surgery.
  The change in ephedrine requirement during surgery (mg).

SECONDARY OUTCOMES:
atropine requirement | every two minutes during surgery
  The change in atropine requirement during surgery (mg).
analgesic requirement | every five minutes during surgery and postoperative 24 hours
  The change in analgesic requirement during surgery and postoperative 24 hours(mg)
blood pressure values | every two minutes during surgery
  The change in systolic and diastolic blood pressure values (mmHg).
heart rate values | every two minutes during surgery
  The change in heart rate values (bpm).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet AKSOY, Assoc.Prof., Principal Investigator — Faculty of Medicine, Ataturk University, Erzurum, Turkey
Locations (1):
- Mehmet AKSOY, Erzurum, string:Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No